CLINICAL TRIAL: NCT06737419
Title: Real World Effectiveness, Persistence, Tolerability, and Safety of Ofatumumab in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS15
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome; Relapsing-remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ofatumumab Cohort: Adult patients diagnosed with MS who started OMB therapy from the time of approval (August 2020).

SUMMARY:
This was a retrospective cohort study using the electronic medical record (EMR) database from Cleveland Clinic. The data was analyzed at start of ofatumumab (OMB) therapy (baseline, defined as 6 months prior to OMB initiation) and at 6 or 12 months following initiation of OMB.

ELIGIBILITY:
Inclusion criteria:

* Patients who initiated OMB commercially from the time of disease modifying therapy (DMT) approval (August 2020), and
* Aged 18 years or older at index date, and
* Patients who met 2017 McDonald Criteria for clinically definite multiple sclerosis (MS), or
* Patients diagnosed with clinically isolated syndrome (CIS) by Cleveland Clinic MS specialist.

Exclusion criteria: Those who were participating in OMB clinical trials (e.g., ARTIOS, OLIKOS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients Categorized by Number of Relapses | Baseline, Month 6, Month 12
Change in Relapse Rate From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12

SECONDARY OUTCOMES:
Age | Baseline
Number of Patients per Demographic Category | Baseline
  Demographics included:
  * Gender
  * Race
  * Ethnicity
Mean Duration of Disease | Baseline
Number of Patients by Most Recent Disease Course | Baseline
  Most recent disease course (in the last 6 months) included relapsing-remitting MS (RRMS)/clinically isolated syndrome (CIS), secondary progressive MS (SPMS), and primary progressive MS (PPMS).
Number of Patients by Patient Determined Disease Steps (PDDS) Score | Baseline, Month 6, Month 12
  The PDDS is a standardized rating scale which is a self-assessment scale of functional disability in MS patients primarily based on ambulation. The questionnaire contained 1 question which was scored ranging from 0 = Normal; 1 = Mild disability; 2 = Moderate disability; 3 = Gait disability; 4 = Early cane; 5 = Late cane; 6 = Bilateral support; and 7 = Wheelchair bound.
Number of Patients Categorized by Comorbidity | Baseline
Number of Patients With no Prior Exposure to Disease Modifying Therapies (DMTs) | Baseline
Number of Prior DMTs | Baseline
Number of Patients who Switched From a DMT to OMB | Baseline
Duration of Time Between Prior DMT and Initiating OMB Treatment | Baseline
Number of Patients by Most Recent Prior DMT | Baseline
  Most recent previous DMTs (in the last 6 months) included high efficacy and medium/low efficacy DMTs.
Number of Patients who Discontinued DMT Prior to OMB Treatment by Reason for Discontinuation | Baseline
Number of Patients by Number of New Brain T2 Lesions | Baseline, Month 6, Month 12
Number of Patients by Number of New Brain Gadolinium Enhancing (GdE) Lesions | Baseline, Month 6, Month 12
Change in Number of New Brain T2 Lesions From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12
Change in Number of New Brain GdE Lesions From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12
Change in PDDS Scores From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12
  The PDDS is a standardized rating scale which is a self-assessment scale of functional disability in MS patients primarily based on ambulation. The questionnaire contained 1 question which was scored ranging from 0 = Normal; 1 = Mild disability; 2 = Moderate disability; 3 = Gait disability; 4 = Early cane; 5 = Late cane; 6 = Bilateral support; and 7 = Wheelchair bound.
Change in Neuro-performance Tests From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12
  Neuro-performance measures included four assessments, cognitive assessment through the processing speed test (PST), upper extremity motor function through the manual dexterity test (MDT), lower extremity function through the walking speed test (WST), and vision assessment through the contrast sensitivity test (CST). PST and CST were scored based on the number of correct responses (with a higher score representing better performance), while MDT and WST were measured based on time to completion (with a lower score representing better performance).
Change in No Evidence of Disease Activity (NEDA) From Baseline to Month 6 and Month 12 After Initiating OMB Treatment | From Baseline up to Month 6 and Month 12
  When available, disability progression measures were calculated for patients. No evidence of disease activity (NEDA-2) status was defined and measured as the absence of clinical relapses and new/enlarging T2 and GdE lesions. NEDA-3 status was defined as components of NEDA-2 and absence of PDDS score worsening. NEDA-2 and NEDA-3 were only evaluated in patients who had all relevant parameters available for review.
Median Change of PDDS From Baseline to Month 6 and Month 12 After Initiation of OMB Treatment | From Baseline up to Month 6 and Month 12
  The PDDS is a standardized rating scale which is a self-assessment scale of functional disability in MS patients primarily based on ambulation. The questionnaire contained 1 question which was scored ranging from 0 = Normal; 1 = Mild disability; 2 = Moderate disability; 3 = Gait disability; 4 = Early cane; 5 = Late cane; 6 = Bilateral support; and 7 = Wheelchair bound.
Number of Patients With 20% or Greater Worsening of Neuro-performance Test Scores After Initiating OMB Treatment | Month 6 and Month 12
  Neuro-performance measures included four assessments, cognitive assessment through the processing speed test (PST), upper extremity motor function through the manual dexterity test (MDT), lower extremity function through the walking speed test (WST), and vision assessment through the contrast sensitivity test (CST). PST and CST were scored based on the number of correct responses (with a higher score representing better performance), while MDT and WST were measured based on time to completion (with a lower score representing better performance).
Number of Patients With 20% or Greater Worsening of PDDS Scores After Initiating OMB Treatment | Month 6 and Month 12
  The PDDS is a standardized rating scale which is a self-assessment scale of functional disability in MS patients primarily based on ambulation. The questionnaire contained 1 question which was scored ranging from 0 = Normal; 1 = Mild disability; 2 = Moderate disability; 3 = Gait disability; 4 = Early cane; 5 = Late cane; 6 = Bilateral support; and 7 = Wheelchair bound.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States